CLINICAL TRIAL: NCT02411123
Title: Prospective Randomized Clinical Study to Evaluate Patient Outcomes Following Pharmacogenetic Testing of Subjects Exhibiting Neuropsychiatric Disorders
Brief Title: Clinical Study to Evaluate Patient Outcomes Following Pharmacogenetic Testing of Subjects Exhibiting Neuropsychiatric Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AltheaDx (Industry)
Collaborators: Carolina Partners in Mental Healthcare (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CLP0002
Record Dates: First submitted 2015-04-01; First posted 2015-04-08 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Depression; Anxiety
Keywords: PGx; pharmacogenetics; depression; anxiety; Neuropsychiatric diseases; IDgenetix; AltheaDx
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDgenetix Neuropsychiatric Test Panel Intervention (Experimental): The medical provider for the IDgenetix Neuropsychiatric Test Panel-guided group will make treatment recommendations based on test results. Patient outcomes will be measured throughout the duration of the study.
  Interventions: Genetic: IDgenetix Neuropsychiatric Test Panel
- control (No Intervention): The medical provider for the control group will not receive IDgenetix Neuropsychiatric Test Panel results and will make treatment recommendations as usual. Patient outcomes will be measured throughout the duration of the study.

INTERVENTIONS:
Genetic: IDgenetix Neuropsychiatric Test Panel — The IDgenetix Neuropsychiatric Test Panel is used to make recommendations on the medication therapy that might be impacted by the genetic background of the patient.
  Other Names: PGx Testing
  Arms: IDgenetix Neuropsychiatric Test Panel Intervention

SUMMARY:
The purpose of this study is to evaluate the effect of pharmacogenetic (PGx) testing on clinical outcomes in a group of subjects exhibiting neuropsychiatric disorders, such as depression and anxiety, as compared to a group of subjects with the same attributes without the guidance of PGx testing for their treatment.

This study will also evaluate whether pharmacogenetic (PGx) testing can reduce adverse drug events, hospitalization rates, hospital length of stay, emergency room visits, disability, death or other serious drug side effects.

DETAILED DESCRIPTION:
Anti-depressant and anti-anxiety medications are still administered by a trial and error method, which results in a substantial number of patients suffering from either a lack of benefit from drug therapy or severe side effects. Approximately 40% of all anti-depressant and anti-anxiety medications prescribed are ineffective, and patients who need to be on medication often discontinue taking their medications, which can have potentially dangerous consequences. Clinical features often fail to predict the drug response and tolerability of a patient to a prescription medication.

Genetics can help guide therapeutic decisions for patients exhibiting neuropsychiatric disorders and improve patient outcomes by maximizing drug efficacy and minimizing the risk of adverse events. Genetics and drug interactions can alter both the pharmacokinetics and pharmacodynamics of a multitude of drug compounds and in turn influence both the safety and efficacy of selected therapeutic regimens.

Pharmacogenetic-guided therapy selection using the IDgenetix Neuropsychiatric Test Panel can enhance patient response and tolerability by facilitating the selection of the most appropriate medication at the most effective dose in the shortest possible time.

In this prospective, randomized, single-blind study, new patients presenting to the clinical site with evidence of depression or anxiety as determined by a qualified clinician will be invited to participate. Study participants will be randomized to one of two groups with respect to the IDgenetix Neuropsychiatric Test Panel result: group with testing results revealed to the medical provider prior to treatment selection (Experimental Group) or group without testing results prior to treatment selection (Control Group). Participant outcomes will be measured at baseline and throughout the 4-month duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18 and 80
* Experiencing or showing evidence of a neuropsychiatric disorder (depression, anxiety, attention deficit hyperactivity disorder and psychosis) as determined by a qualified clinician
* Subjects new to the medical provider
* Willing and able to comply with study procedures
* Able to provide written informed consent

Exclusion Criteria:

* Unwilling or unable to provide written informed consent and to comply with study procedures
* Any subject for whom providing a buccal swab sample would be contraindicated or not possible
* Subject with a history of chronic renal dysfunction, Chronic Kidney Disease (Stage 4 or 5)
* Abnormal hepatic function within the last 2 years (INR >1.2 not attributable to anticoagulant medications, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5x normal, or suspected cirrhosis
* History of malabsorption (short gut syndrome)
* Any gastric or small bowel surgery less than 3 months prior to study enrollment
* Subject is being treated with intravenous medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Comparison of change in neuropsychiatric state between the two treatment arms measured by Neuropsychiatric Questionnaire (NPQ) | 4 months
  Neuropsychiatric Questionnaire (NPQ) score change comparison between the two treatment arms over a 4-month period.
Comparison of change in responsiveness between the two treatment arms measured by Symbol Digit Coding (SDC) test | 4 months
  Symbol Digit Coding (SDC) test score change comparison between the two treatment arms over a 4-month period.

SECONDARY OUTCOMES:
Comparison of hospital utilization between the two treatment arms as measured by hospital admission and re-admission rates | 4 months
  Comparison of hospital utilization, as measured by hospital admission and re-admission rates, between the two treatment arms over a 4-month period.
Comparison of adverse drug events between the two treatment arms over a 4-month period | 4 months
  Comparison of adverse drug events between the two treatment arms over a 4-month period

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina Partners in Mental HealthCare, Raleigh, North Carolina, United States

REFERENCES:
- [Background] Masand PS. Tolerability and adherence issues in antidepressant therapy. Clin Ther. 2003 Aug;25(8):2289-304. doi: 10.1016/s0149-2918(03)80220-5. PMID 14512135
- [Background] Crisafulli C, Fabbri C, Porcelli S, Drago A, Spina E, De Ronchi D, Serretti A. Pharmacogenetics of antidepressants. Front Pharmacol. 2011 Feb 16;2:6. doi: 10.3389/fphar.2011.00006. eCollection 2011. PMID 21687501
- [Background] Mrazek DA. Psychiatric pharmacogenomic testing in clinical practice. Dialogues Clin Neurosci. 2010;12(1):69-76. doi: 10.31887/DCNS.2010.12.1/dmrazek. PMID 20373668
- [Background] Serretti A, Kato M, De Ronchi D, Kinoshita T. Meta-analysis of serotonin transporter gene promoter polymorphism (5-HTTLPR) association with selective serotonin reuptake inhibitor efficacy in depressed patients. Mol Psychiatry. 2007 Mar;12(3):247-57. doi: 10.1038/sj.mp.4001926. Epub 2006 Dec 5. PMID 17146470
- [Derived] Olson MC, Maciel A, Gariepy JF, Cullors A, Saldivar JS, Taylor D, Centeno J, Garces JA, Vaishnavi S. Clinical Impact of Pharmacogenetic-Guided Treatment for Patients Exhibiting Neuropsychiatric Disorders: A Randomized Controlled Trial. Prim Care Companion CNS Disord. 2017 Mar 16;19(2). doi: 10.4088/PCC.16m02036. PMID 28314093